CLINICAL TRIAL: NCT00594646
Title: A Phase IV Open-Label Evaluation of Safety, Tolerability and Patient Acceptance of Raltegravir (MK-0518) Combined With a Fixed-Dose Formulation of Tenofovir Following Potential Exposure to HIV-1
Brief Title: HIV Non Occupational Post-Exposure Prophylaxis (PEP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fenway Community Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kenneth H. Mayer, MD, Medical Director, The Fenway Institute, Fenway Community Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MK PEP 2007
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: HIV Infections
Keywords: HIV Prevention; Non-occupational post-exposure prophylaxis; HIV seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Raltegravir Potassium; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (Other): TRUVADA
  Interventions: Drug: TRUVADA + Raltegravir

INTERVENTIONS:
Drug: TRUVADA + Raltegravir — TRUVADA (tenofovir disoproxil fumarate (DF) 300mg + emtricitabine 200mg) + RALTEGRAVIR 400mg
  Other Names: tenofovir DF; emtricitabine

SUMMARY:
This study will evaluate how safe and tolerable a combination of taking three-drugs will be for the purpose of preventing HIV transmission after a high-risk sexual contact exposure in HIV uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate a three drug regimen in the form of two pills which will be taken for 28 days for the prevention of HIV infection. Two drugs are combined in an FDA-approved pill called TRUVADA, containing the HIV medications, tenofovir disoproxil fumarate 300mg and emtricitabine 200mg, taken as one pill once a day. The third drug is a new formulation, raltegravir 400mg pill taken twice a day.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected on the basis of a negative HIV Rapid Test, EIA or Western blot, and a negative HIV-1 RNA assay
* Possible non-occupational exposure to HIV-1, recent enough to permit receiving the first dose of study medication within 72 hours from the end of the exposure.
* Able to understand the study procedures and willing to sign informed consent

Exclusion Criteria:

* Any active psychiatric illness or active drug or alcohol abuse that, in the opinion of the investigator, could prevent compliance with study procedures.
* Pregnancy.
* Chronic hepatitis B infection, diagnosed by either positive serum HBsAg or positive serum HBV DNA; or prior lamivudine therapy for hepatitis B.
* Creatinine clearance less than 50 mL/min as calculated by Cockcroft-Gault formula.
* Unwillingness to participate in study procedures, including Mental Health referral and intervention.
* Known intolerance or allergy to tenofovir DF, emtricitabine or raltegravir.
* Use of prohibited concomitant medication: dilantin, phenobarbital and rifampin which cannot be used with raltegravir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Mayer, MD, Principal Investigator — Fenway Community Health
Locations (1):
- Fenway Community Health, Boston, Massachusetts, United States

REFERENCES:
- [Result] Mayer KH, Mimiaga MJ, Gelman M, Grasso C. Raltegravir, tenofovir DF, and emtricitabine for postexposure prophylaxis to prevent the sexual transmission of HIV: safety, tolerability, and adherence. J Acquir Immune Defic Syndr. 2012 Apr 1;59(4):354-9. doi: 10.1097/QAI.0b013e31824a03b8. PMID 22267017
- See also: Link to full-text publication — http://journals.lww.com/jaids/Fulltext/2012/04010/Raltegravir,_Tenofovir_DF,_and_Emtricitabine_for.6.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Fenway Health. Patients at least 18 years of age, who contacted Fenway Health and presented within 72 hours after a potential sexual exposure to HIV-1 were asked to participate in this study.
Pre-assignment Details: If study coordinator is notified more than 72 hours after exposure occurred, person will not be eligible for study participation; however they will be referred to an on call medical provider for Non Occupational Post-Exposure Prophylaxis evaluation.
Groups:
- TRUVADA + Raltegravir: Men or women, 18 years of age or older, who present within 72 hours of a potential non-occupational exposure to HIV-1.
Period: Overall Study
Arm/Group | TRUVADA + Raltegravir
Started | 100
Completed | 84
Not Completed | 16
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 15

BASELINE CHARACTERISTICS:
Groups:
- Group 1: TRUVADA (tenofovir DF 300mg + emtricitabine 200mg) + raltegravir (400mg)
Arm/Group | Group 1
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 100
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 33.3 [18 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 11
  White | 71
  More than one race | 13
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Medication Regimen Completion Rates
Description: Pill counts performed at 14 and 28 days
Time Frame: 28 days
Measure: Number; unit: participants
Groups:
- Group 1: TDF 300mg + FTC 200mg (TDF/FTC) once daily + raltegravir 400mg twice daily
Arm/Group | Group 1
Number analyzed (Participants) | 100
participants
  Completed as prescribed | 57
  Stopped or Modified regimen | 28
  Lost to follow-up | 15

2. Primary Outcome: Number of HIV-1 Infected Participants
Description: Of participants that were evaluable at 3 months post initiation of treatment, how many became HIV-1 infected
Time Frame: 90 days
Population: Participants evaluable at 3 months (90 days) after treatment initiation
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 85
participants | 0

ADVERSE EVENTS:
Time Frame: 28 days
Groups:
- Group 1: TDF 300mg and FTC 200mg (TDF/FTC) once daily + raltegravir (400mg) twice daily
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 93/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=100)
Diarrhea / Loose Stool / Soft Stool (Gastrointestinal disorders) | 21
Fatigue (General disorders) | 14
Abdominal discomfort, pain, gas, or bloating (Gastrointestinal disorders) | 16
Nausea/vomiting (Gastrointestinal disorders) | 27
Headache (Nervous system disorders) | 15

LIMITATIONS AND CAVEATS:
Limitations of the current study included:

1. Reliance on self-reports to measure adherence
2. Study population almost exclusively male (reflecting the demographics of people who call Fenway Health's hotline after an acute sexual exposure)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No